CLINICAL TRIAL: NCT04034004
Title: The Role of Endogenous Opioids in Mindfulness-based Chronic Pain Relief
Brief Title: Chronic Low Back Pain and Meditation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Fadel Zeidan, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 190709; R21AT010352 (NIH)
Record Dates: First submitted 2019-05-09; First posted 2019-07-26 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Pain
Keywords: Mindfulness; Opioids; Pain; Naloxone
MeSH Terms: conditions — Pain | interventions — Mindfulness; Naloxone; Sodium Chloride; Meditation

STUDY DESIGN:
Intervention Model Description: The study will employ a double blinded crossover factorial design. Baseline pain ratings will be assessed using visual analog scales obtained during three sessions where low back pain is induced. Study volunteers will participate in a four session (20min/session) meditation intervention. After meditation training, subjects will report to the UCSD Altman Clinical and Translational Research Institute across two separate experimental sessions. Half of the volunteers will be administered naloxone (opioid antagonist; 0.15 mg/kg bolus+ 0.1 mg/kg/hour infusion) and the other in the subsequent session will be administered IV placebo-saline, vice versa.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the study physician, research coordinator, and research pharmacist will be aware of drug assignments. Research staff (nurses; research technicians) and the PI will be blinded to drug assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Meditation (Experimental): Subjects will participate in four sessions (20 min/session) of mindfulness training. Participants will be taught that perceived sensory events are "momentary" and "fleeting" and require no further evaluation.
  Interventions: Behavioral: Mindfulness; Drug: Naloxone; Other: Saline; Behavioral: Meditation
- meditation (Experimental): Subjects will participate in four sessions (20 min/session) of mindfulness training. Participants will be taught that perceived sensory events are "momentary" and "fleeting" and require no further evaluation.
  Interventions: Behavioral: Mindfulness; Drug: Naloxone; Other: Saline; Behavioral: Meditation

INTERVENTIONS:
Behavioral: Mindfulness — A well-validated brief meditation-based mental training regimen [four sessions; 20 min/session] is used to teach patients to independently practice closing their eyes and take a deep breath every few minutes.
  Other Names: mental training
Drug: Naloxone — A 0.15 mg/kg bolus dose of naloxone (Naloxone hydrochloride, Amphastar Pharmaceuticals, Inc., Rancho Cucamonga, California) in 25ml normal saline will be administered over 10 minutes. The investigators also will administer a supplementary IV infusion dose of 0.1mg/kg/hour naloxone immediately after bolus infusion will cease till the end of the experiment.
Other: Saline — A 0.15 mg/kg bolus dose of saline in 25ml normal saline will be administered over 10 minutes. The investigators also will administer a supplementary IV infusion dose of 0.1mg/kg/hour saline immediately after bolus infusion will cease till the end of the experiment.
Behavioral: Meditation — A well-validated brief meditation-based mental training regimen [four sessions; 20 min/session] is used to teach patients to independently practice closing their eyes and take a deep breath every few minutes.
  Other Names: mental training

SUMMARY:
The purpose of this research study is to see if and how mindfulness meditation affects pain. Specifically, we are interested in assessing if mindfulness is associated with the release of naturally occurring opiates in the body, in response to intravenous (IV) administration of the opioid antagonist naloxone during a chronic low back pain provoking procedure.

DETAILED DESCRIPTION:
The purpose of this psychophysical and pharmacologic study is to determine if meditation induced pain relief is mediated by endogenous opioids in response to intravenous (IV) administration of the opioid antagonist naloxone during a pain evoking straight leg raise test in response to double-blind intravenous administration (IV) of naloxone/placebo-saline. The aim of this study is to determine if mindfulness-based analgesia is associated with the release of endogenous opioids.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a medical evaluation that demonstrates chronic low back pain that is evoked by lifting the legs. Existing medical records, per physician discretion and low back examinations will confirm diagnosis
* Participants must be between 18 and 65 years of age
* Participants must rate their daily chronic pain intensity at a 3 or higher on 0-10 visual analog scale
* Participants must have experienced their chronic low back pain for at least 3 months
* Participants must have no prior meditative experience
* Participants must be straight leg raise test positive

Exclusion Criteria:

* Participants must not be participating in any new (within 2 weeks prior or anytime after enrollment) pain management procedures during the study period
* Participants must not be taking opioids
* Participants must not be pregnant or nursing mothers
* Participants must have not had back surgery within the last year before their enrollment into the study
* Participants must have not had any other sensory or motor deficits that preclude participation in this study
* Participants must not have known anomalies of the central nervous system including: stroke, dementia, aneurysm, and a personal history of psychosis
* Participants must not have any known allergies to naloxone or similar drugs
* Participants must not have a history of syncope and/or fear of needles/blood

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fadel Zeidan, PhD, Principal Investigator — UC San Diego
Locations (2):
- United States (2):
  - Altman Clinical and Translational Research Institute, La Jolla, California
  - UC San Diego Center for Mindfulness, San Diego, California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Anderson WS, Sheth RN, Bencherif B, Frost JJ, Campbell JN. Naloxone increases pain induced by topical capsaicin in healthy human volunteers. Pain. 2002 Sep;99(1-2):207-16. doi: 10.1016/s0304-3959(02)00103-3. PMID 12237198
- [Background] Andersson GB. Epidemiological features of chronic low-back pain. Lancet. 1999 Aug 14;354(9178):581-5. doi: 10.1016/S0140-6736(99)01312-4. PMID 10470716
- [Background] Apkarian AV, Krauss BR, Fredrickson BE, Szeverenyi NM. Imaging the pain of low back pain: functional magnetic resonance imaging in combination with monitoring subjective pain perception allows the study of clinical pain states. Neurosci Lett. 2001 Feb 16;299(1-2):57-60. doi: 10.1016/s0304-3940(01)01504-x. PMID 11166937
- [Background] Bencherif B, Fuchs PN, Sheth R, Dannals RF, Campbell JN, Frost JJ. Pain activation of human supraspinal opioid pathways as demonstrated by [11C]-carfentanil and positron emission tomography (PET). Pain. 2002 Oct;99(3):589-598. doi: 10.1016/S0304-3959(02)00266-X. PMID 12406535
- [Background] Brown CA, Matthews J, Fairclough M, McMahon A, Barnett E, Al-Kaysi A, El-Deredy W, Jones AKP. Striatal opioid receptor availability is related to acute and chronic pain perception in arthritis: does opioid adaptation increase resilience to chronic pain? Pain. 2015 Nov;156(11):2267-2275. doi: 10.1097/j.pain.0000000000000299. PMID 26176892
- [Background] Bruehl S, Burns JW, Passik SD, Gupta R, Buvanendran A, Chont M, Schuster E, Orlowska D, France CR. The Contribution of Differential Opioid Responsiveness to Identification of Opioid Risk in Chronic Pain Patients. J Pain. 2015 Jul;16(7):666-75. doi: 10.1016/j.jpain.2015.04.001. Epub 2015 Apr 16. PMID 25892658
- [Background] Bruehl S, Chung OY. Parental history of chronic pain may be associated with impairments in endogenous opioid analgesic systems. Pain. 2006 Oct;124(3):287-294. doi: 10.1016/j.pain.2006.04.018. Epub 2006 May 24. PMID 16725261
- [Background] Bruehl S, Chung OY, Burns JW, Biridepalli S. The association between anger expression and chronic pain intensity: evidence for partial mediation by endogenous opioid dysfunction. Pain. 2003 Dec;106(3):317-324. doi: 10.1016/S0304-3959(03)00319-1. PMID 14659514
- [Background] Bruehl S, Chung OY, Burns JW, Diedrich L. Trait anger expressiveness and pain-induced beta-endorphin release: support for the opioid dysfunction hypothesis. Pain. 2007 Aug;130(3):208-215. doi: 10.1016/j.pain.2006.11.013. Epub 2007 Jan 2. PMID 17197088
- [Background] Bruno PA, Millar DP, Goertzen DA. Inter-rater agreement, sensitivity, and specificity of the prone hip extension test and active straight leg raise test. Chiropr Man Therap. 2014 Jun 16;22:23. doi: 10.1186/2045-709X-22-23. eCollection 2014. PMID 24982755
- [Background] Burns JW, Bruehl S, France CR, Schuster E, Orlowska D, Chont M, Gupta RK, Buvanendran A. Endogenous Opioid Function and Responses to Morphine: The Moderating Effects of Anger Expressiveness. J Pain. 2017 Aug;18(8):923-932. doi: 10.1016/j.jpain.2017.02.439. Epub 2017 Mar 30. PMID 28365372
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, DeLitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH Task Force on Research Standards for Chronic Low Back Pain. Int J Ther Massage Bodywork. 2015 Sep 1;8(3):16-33. doi: 10.3822/ijtmb.v8i3.295. eCollection 2015 Sep. PMID 26388962
- [Background] Deyo RA, Mirza SK, Turner JA, Martin BI. Overtreating chronic back pain: time to back off? J Am Board Fam Med. 2009 Jan-Feb;22(1):62-8. doi: 10.3122/jabfm.2009.01.080102. PMID 19124635
- [Background] DosSantos MF, Martikainen IK, Nascimento TD, Love TM, Deboer MD, Maslowski EC, Monteiro AA, Vincent MB, Zubieta JK, DaSilva AF. Reduced basal ganglia mu-opioid receptor availability in trigeminal neuropathic pain: a pilot study. Mol Pain. 2012 Sep 24;8:74. doi: 10.1186/1744-8069-8-74. PMID 23006894
- [Background] Fardon DF. Nomenclature and classification of lumbar disc pathology. Spine (Phila Pa 1976). 2001 Mar 1;26(5):461-2. doi: 10.1097/00007632-200103010-00007. No abstract available. PMID 11242371
- [Background] Fardon DF, Williams AL, Dohring EJ, Murtagh FR, Gabriel Rothman SL, Sze GK. Lumbar disc nomenclature: version 2.0: Recommendations of the combined task forces of the North American Spine Society, the American Society of Spine Radiology and the American Society of Neuroradiology. Spine J. 2014 Nov 1;14(11):2525-45. doi: 10.1016/j.spinee.2014.04.022. Epub 2014 Apr 24. PMID 24768732
- [Background] Han B, Compton WM, Jones CM, Cai R. Nonmedical Prescription Opioid Use and Use Disorders Among Adults Aged 18 Through 64 Years in the United States, 2003-2013. JAMA. 2015 Oct 13;314(14):1468-78. doi: 10.1001/jama.2015.11859. PMID 26461997
- [Background] Harris RE, Clauw DJ, Scott DJ, McLean SA, Gracely RH, Zubieta JK. Decreased central mu-opioid receptor availability in fibromyalgia. J Neurosci. 2007 Sep 12;27(37):10000-6. doi: 10.1523/JNEUROSCI.2849-07.2007. PMID 17855614
- [Background] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424
- [Background] Institute of Medicine (US) Committee on Advancing Pain Research, Care, and Education. Relieving Pain in America: A Blueprint for Transforming Prevention, Care, Education, and Research. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK91497/ PMID 22553896
- [Background] Jacob JA. As Opioid Prescribing Guidelines Tighten, Mindfulness Meditation Holds Promise for Pain Relief. JAMA. 2016 Jun 14;315(22):2385-7. doi: 10.1001/jama.2016.4875. No abstract available. PMID 27203730
- [Background] Jamison RN, Ross EL, Michna E, Chen LQ, Holcomb C, Wasan AD. Substance misuse treatment for high-risk chronic pain patients on opioid therapy: a randomized trial. Pain. 2010 Sep;150(3):390-400. doi: 10.1016/j.pain.2010.02.033. Epub 2010 Mar 23. PMID 20334973
- [Background] Jones AK, Cunningham VJ, Ha-Kawa S, Fujiwara T, Luthra SK, Silva S, Derbyshire S, Jones T. Changes in central opioid receptor binding in relation to inflammation and pain in patients with rheumatoid arthritis. Br J Rheumatol. 1994 Oct;33(10):909-16. doi: 10.1093/rheumatology/33.10.909. PMID 7921749
- [Background] Jones AK, Kitchen ND, Watabe H, Cunningham VJ, Jones T, Luthra SK, Thomas DG. Measurement of changes in opioid receptor binding in vivo during trigeminal neuralgic pain using [11C] diprenorphine and positron emission tomography. J Cereb Blood Flow Metab. 1999 Jul;19(7):803-8. doi: 10.1097/00004647-199907000-00011. PMID 10413036
- [Background] Jones AK, Watabe H, Cunningham VJ, Jones T. Cerebral decreases in opioid receptor binding in patients with central neuropathic pain measured by [11C]diprenorphine binding and PET. Eur J Pain. 2004 Oct;8(5):479-85. doi: 10.1016/j.ejpain.2003.11.017. PMID 15324779
- [Background] Klega A, Eberle T, Buchholz HG, Maus S, Maihofner C, Schreckenberger M, Birklein F. Central opioidergic neurotransmission in complex regional pain syndrome. Neurology. 2010 Jul 13;75(2):129-36. doi: 10.1212/WNL.0b013e3181e7ca2e. PMID 20625165
- [Background] Kwong EH, Virani N, Robert M, Gerry K, Harding A, Rose MS, Dukelow SP, Barton PM. Inter-rater reliability of the Active Straight-Leg Raise and One-Leg Standing tests in non-pregnant women. J Rehabil Med. 2013 Nov;45(10):1058-64. doi: 10.2340/16501977-1213. PMID 23995959
- [Background] Loggia ML, Kim J, Gollub RL, Vangel MG, Kirsch I, Kong J, Wasan AD, Napadow V. Default mode network connectivity encodes clinical pain: an arterial spin labeling study. Pain. 2013 Jan;154(1):24-33. doi: 10.1016/j.pain.2012.07.029. Epub 2012 Oct 27. PMID 23111164
- [Background] Maarrawi J, Peyron R, Mertens P, Costes N, Magnin M, Sindou M, Laurent B, Garcia-Larrea L. Differential brain opioid receptor availability in central and peripheral neuropathic pain. Pain. 2007 Jan;127(1-2):183-94. doi: 10.1016/j.pain.2006.10.013. Epub 2006 Nov 29. PMID 17137714
- [Background] Martikainen IK, Pecina M, Love TM, Nuechterlein EB, Cummiford CM, Green CR, Harris RE, Stohler CS, Zubieta JK. Alterations in endogenous opioid functional measures in chronic back pain. J Neurosci. 2013 Sep 11;33(37):14729-37. doi: 10.1523/JNEUROSCI.1400-13.2013. PMID 24027273
- [Background] May LM, Kosek P, Zeidan F, Berkman ET. Enhancement of Meditation Analgesia by Opioid Antagonist in Experienced Meditators. Psychosom Med. 2018 Nov/Dec;80(9):807-813. doi: 10.1097/PSY.0000000000000580. PMID 29595707
- [Background] Mens JM, Vleeming A, Snijders CJ, Stam HJ, Ginai AZ. The active straight leg raising test and mobility of the pelvic joints. Eur Spine J. 1999;8(6):468-73. doi: 10.1007/s005860050206. PMID 10664304
- [Background] Nelson LS, Juurlink DN, Perrone J. Addressing the Opioid Epidemic. JAMA. 2015 Oct 13;314(14):1453-4. doi: 10.1001/jama.2015.12397. No abstract available. PMID 26461995
- [Background] Ngai SH, Berkowitz BA, Yang JC, Hempstead J, Spector S. Pharmacokinetics of naloxone in rats and in man: basis for its potency and short duration of action. Anesthesiology. 1976 May;44(5):398-401. doi: 10.1097/00000542-197605000-00008. PMID 1267205
- [Background] Rebain R, Baxter GD, McDonough S. A systematic review of the passive straight leg raising test as a diagnostic aid for low back pain (1989 to 2000). Spine (Phila Pa 1976). 2002 Sep 1;27(17):E388-95. doi: 10.1097/00007632-200209010-00025. PMID 12221373
- [Background] Roussel NA, Nijs J, Truijen S, Smeuninx L, Stassijns G. Low back pain: clinimetric properties of the Trendelenburg test, active straight leg raise test, and breathing pattern during active straight leg raising. J Manipulative Physiol Ther. 2007 May;30(4):270-8. doi: 10.1016/j.jmpt.2007.03.001. PMID 17509436
- [Background] Saloner B, Karthikeyan S. Changes in Substance Abuse Treatment Use Among Individuals With Opioid Use Disorders in the United States, 2004-2013. JAMA. 2015 Oct 13;314(14):1515-7. doi: 10.1001/jama.2015.10345. No abstract available. PMID 26462001
- [Background] Sharma HA, Gupta R, Olivero W. fMRI in patients with lumbar disc disease: a paradigm to study patients over time. J Pain Res. 2011;4:401-5. doi: 10.2147/JPR.S24393. Epub 2011 Dec 7. PMID 22247623
- [Background] Steglitz J, Buscemi J, Ferguson MJ. The future of pain research, education, and treatment: a summary of the IOM report "Relieving pain in America: a blueprint for transforming prevention, care, education, and research". Transl Behav Med. 2012 Mar;2(1):6-8. doi: 10.1007/s13142-012-0110-2. PMID 24073092
- [Background] Summers B, Malhan K, Cassar-Pullicino V. Low back pain on passive straight leg raising: the anterior theca as a source of pain. Spine (Phila Pa 1976). 2005 Feb 1;30(3):342-5. doi: 10.1097/01.brs.0000152378.93868.c8. PMID 15682017
- [Background] Thompson SJ, Pitcher MH, Stone LS, Tarum F, Niu G, Chen X, Kiesewetter DO, Schweinhardt P, Bushnell MC. Chronic neuropathic pain reduces opioid receptor availability with associated anhedonia in rat. Pain. 2018 Sep;159(9):1856-1866. doi: 10.1097/j.pain.0000000000001282. PMID 29794614
- [Background] Wasan AD, Davar G, Jamison R. The association between negative affect and opioid analgesia in patients with discogenic low back pain. Pain. 2005 Oct;117(3):450-461. doi: 10.1016/j.pain.2005.08.006. PMID 16154274
- [Background] Wasan AD, Loggia ML, Chen LQ, Napadow V, Kong J, Gollub RL. Neural correlates of chronic low back pain measured by arterial spin labeling. Anesthesiology. 2011 Aug;115(2):364-74. doi: 10.1097/ALN.0b013e318220e880. PMID 21720241
- [Background] Zeidan F, Adler-Neal AL, Wells RE, Stagnaro E, May LM, Eisenach JC, McHaffie JG, Coghill RC. Mindfulness-Meditation-Based Pain Relief Is Not Mediated by Endogenous Opioids. J Neurosci. 2016 Mar 16;36(11):3391-7. doi: 10.1523/JNEUROSCI.4328-15.2016. PMID 26985045
- [Background] Zeidan F, Emerson NM, Farris SR, Ray JN, Jung Y, McHaffie JG, Coghill RC. Mindfulness Meditation-Based Pain Relief Employs Different Neural Mechanisms Than Placebo and Sham Mindfulness Meditation-Induced Analgesia. J Neurosci. 2015 Nov 18;35(46):15307-25. doi: 10.1523/JNEUROSCI.2542-15.2015. PMID 26586819
- [Background] Zeidan F, Gordon NS, Merchant J, Goolkasian P. The effects of brief mindfulness meditation training on experimentally induced pain. J Pain. 2010 Mar;11(3):199-209. doi: 10.1016/j.jpain.2009.07.015. Epub 2009 Oct 22. PMID 19853530
- [Background] Zeidan F, Grant JA, Brown CA, McHaffie JG, Coghill RC. Mindfulness meditation-related pain relief: evidence for unique brain mechanisms in the regulation of pain. Neurosci Lett. 2012 Jun 29;520(2):165-73. doi: 10.1016/j.neulet.2012.03.082. Epub 2012 Apr 6. PMID 22487846
- [Background] Zeidan F, Johnson SK, Diamond BJ, David Z, Goolkasian P. Mindfulness meditation improves cognition: evidence of brief mental training. Conscious Cogn. 2010 Jun;19(2):597-605. doi: 10.1016/j.concog.2010.03.014. Epub 2010 Apr 3. PMID 20363650
- [Background] Zeidan F, Johnson SK, Gordon NS, Goolkasian P. Effects of brief and sham mindfulness meditation on mood and cardiovascular variables. J Altern Complement Med. 2010 Aug;16(8):867-73. doi: 10.1089/acm.2009.0321. PMID 20666590
- [Background] Zeidan F, Lobanov OV, Kraft RA, Coghill RC. Brain mechanisms supporting violated expectations of pain. Pain. 2015 Sep;156(9):1772-1785. doi: 10.1097/j.pain.0000000000000231. PMID 26083664
- [Background] Zeidan F, Martucci KT, Kraft RA, Gordon NS, McHaffie JG, Coghill RC. Brain mechanisms supporting the modulation of pain by mindfulness meditation. J Neurosci. 2011 Apr 6;31(14):5540-8. doi: 10.1523/JNEUROSCI.5791-10.2011. PMID 21471390
- [Background] Zeidan F, Martucci KT, Kraft RA, McHaffie JG, Coghill RC. Neural correlates of mindfulness meditation-related anxiety relief. Soc Cogn Affect Neurosci. 2014 Jun;9(6):751-9. doi: 10.1093/scan/nst041. Epub 2013 Apr 24. PMID 23615765
- [Background] Zubieta JK, Smith YR, Bueller JA, Xu Y, Kilbourn MR, Jewett DM, Meyer CR, Koeppe RA, Stohler CS. Regional mu opioid receptor regulation of sensory and affective dimensions of pain. Science. 2001 Jul 13;293(5528):311-5. doi: 10.1126/science.1060952. PMID 11452128
- [Background] Zubieta JK, Smith YR, Bueller JA, Xu Y, Kilbourn MR, Jewett DM, Meyer CR, Koeppe RA, Stohler CS. mu-opioid receptor-mediated antinociceptive responses differ in men and women. J Neurosci. 2002 Jun 15;22(12):5100-7. doi: 10.1523/JNEUROSCI.22-12-05100.2002. PMID 12077205
- [Derived] Khatib L, Dean JG, Oliva V, Riegner G, Gonzalez NE, Birenbaum J, Cruanes GF, Miller J, Patterson M, Kim HC, Chakravarthy K, Zeidan F. The role of endogenous opioids in mindfulness and sham mindfulness-meditation for the direct alleviation of evoked chronic low back pain: a randomized clinical trial. Neuropsychopharmacology. 2024 Jun;49(7):1069-1077. doi: 10.1038/s41386-023-01766-2. Epub 2023 Nov 20. PMID 37985872

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 500 individuals were screened for eligibility through the UCSD Recruitment services and study flyers. Enrollment started in January 2021 and data collection was completed in December of 2022.
Pre-assignment Details: 88 out of the 500 individuals were enrolled and participated in the baseline session. Seventeen out of the 88 were not randomized for the following reasons: Not responsive to straight leg raise test (n = 4), Intolerance to pain procedures (n = 3), Withdrew (n = 3), Scheduling issues (n = 1), Transportation issues (n = 1), Positive opioid test (n = 1), Inappropriate behavior (n = 1), Other pain management (n = 1), instruction incomprehension (n = 1) and Mindfulness experience (n = 1).
Groups:
- Mindfulness Meditation and Saline First: After providing informed consent, 18 participants completed baseline testing.
  Participants then completed a four session mindfulness meditation intervention where participants were taught that perceived sensory events are "momentary" and "fleeting" and require no further evaluation. One participant dropped out after the first intervention session.
  After their respective intervention, these participants received IV saline in session 6. Two participants were dismissed because of trouble administering the IV.
  Saline: A 0.15 mg/kg bolus dose of saline in 25ml normal saline will be administered over 10 minutes. The investigators also will administer a supplementary IV infusion dose of 0.1mg/kg/hour saline immediately after bolus infusion will cease till the end of the experiment.
  After a two day washout period, 15 participants returned to the clinic and performed the naloxone infusion in session 7.
  Naloxone: A 0.15 mg/kg bolus dose of naloxone (Naloxone hydrochloride, Amphastar Pharmaceuticals, Inc., Rancho Cucamonga, California) in 25ml normal saline will be administered over 10 minutes. The investigators also administered a supplementary IV infusion dose of 0.1mg/kg/hour naloxone immediately after bolus infusion will cease till the end of the experiment.
- Non Mindfulness Meditation and Saline First: After providing informed consent, 18 participants completed baseline testing. 2 participants withdrew from this session
  Participants then completed a four session non-mindfulness meditation intervention where participants were taught to independently practice closing their eyes and take a deep breath every few minutes.
  After their respective intervention, these participants received IV saline in session 6. One participants was dismissed because of trouble administering the IV.
  After a two day washout period, 15 participants returned to the clinic and performed the naloxone infusion in session 7.
- Mindfulness Meditation and Naloxone First: After providing informed consent, 17 participants participated in baseline testing. Two participants withdrew for scheduling issues after baseline.
  Fifteen participants then completed a four session mindfulness meditation intervention where they were taught to focus on the changing sensations of the breath non-reactively
  After their respective intervention, these 15 participants received IV naloxone in session 6
  After a two day washout period, 15 participants returned to the clinic and performed the saline infusion in session 7.
- Non Mindfulness Meditation and Naloxone First: After providing informed consent, 18 participants participated in baseline testing. Three participants withdrew for scheduling issues after baseline.
  Fifteen participants then completed a four session non mindfulness meditation intervention where they were taught to independently take deep breaths.
  After their respective intervention, these participants received IV naloxone in session 6. However, a study nurse unintentionally instructed a patient that naloxone was to be infused and thus the participant was dismissed.
  After a two day washout period, 14 participants returned to the clinic and performed the saline infusion in session 7.
Period: Overall Study
Arm/Group | Mindfulness Meditation and Saline First | Non Mindfulness Meditation and Saline First | Mindfulness Meditation and Naloxone First | Non Mindfulness Meditation and Naloxone First
Started | 18 | 18 | 17 | 18
Completed | 15 | 15 | 15 | 14
Not Completed | 3 | 3 | 2 | 4
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 3
Not completed — could not find vein to administer IV | 2 | 1 | 0 | 0
Not completed — nurse accidentally unblinded subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population was not different from the assignment in participant flow.
Groups:
- Mindfulness Meditation; Non-mindfulness Meditation: Subjects will participate in four sessions (20 min/session) of mindfulness training. Participants will be taught that perceived sensory events are "momentary" and "fleeting" and require no further evaluation.
  Mindfulness: A well-validated brief meditation-based mental training regimen [four sessions; 20 min/session] is used to teach patients to independently practice closing their eyes and take a deep breath every few minutes.
  Naloxone: A 0.15 mg/kg bolus dose of naloxone (Naloxone hydrochloride, Amphastar Pharmaceuticals, Inc., Rancho Cucamonga, California) in 25ml normal saline will be administered over 10 minutes. The investigators also will administer a supplementary IV infusion dose of 0.1mg/kg/hour naloxone immediately after bolus infusion will cease till the end of the experiment.
  Saline: A 0.15 mg/kg bolus dose of saline in 25ml normal saline will be administered over 10 minutes. The investigators also will administer a supplementary IV infusion dose of 0.1mg/kg/hour saline immediately after bolus infusion will cease till the end of the experiment.
  Meditation: A well-validated brief meditation-based mental training regimen [four sessions; 20 min/session] is used to teach patients to independently practice closing their eyes and take a deep breath every few minutes.
- Total: Total of all reporting groups
Arm/Group | Mindfulness Meditation | Non-mindfulness Meditation | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years]
  age | 45 (12) | 47 (13) | 46 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 15 | 14 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 26 | 19 | 45
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0
Numerical pain ratings [Mean (Standard Deviation); unit: units on a scale] — Straight leg raise test induced numerical pain ratings were assessed using an 11-point scale where the minimum rating ("0") was designated as "no pain sensation" and the maximum ("10") as "most intense pain imaginable".
  Pain ratings were collected while patients were lying on backs and in response to the straight leg raise test (SLR).
  The following ratings correspond to the first SLR in the baseline session. Higher numerical ratings equated to higher pain.
  units on a scale
    straight leg raise test | 4.83 (2.21) | 5.41 (2.46) | 5.12 (2.34)
    supine | 3.60 (2.08) | 4.69 (2.25) | 4.14 (2.22)

OUTCOME MEASURES:

1. Primary Outcome: Pain Ratings
Description: Numerical pain ratings (NRS) will be assessed while lying on the back and in response to the straight leg raise test (SLR). Pain ratings will be collected during SLR 1 and SLR 2 in the baseline, saline and naloxone sessions, respectively. The 11 point scan will include a minimum rating of "0" which is characterized as "no pain" whereas the maximum ("10") is labeled as "most intense imaginable"." Higher numbers correspond to higher pain.
Time Frame: Pain ratings were collected while lying supine and in response to the straight leg raise test. Collected twice, once in the first half and one in the second half of the baseline, saline infusion and naloxone infusion sessions. Up to 8 weeks total.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Non Mindfulness Meditation: Subjects will participate in four sessions (20 min/session) of mindfulness training. Participants will be taught that perceived sensory events are "momentary" and "fleeting" and require no further evaluation.
  Mindfulness: A well-validated brief meditation-based mental training regimen [four sessions; 20 min/session] is used to teach patients to independently practice closing their eyes and take a deep breath every few minutes.
  Naloxone: A 0.15 mg/kg bolus dose of naloxone (Naloxone hydrochloride, Amphastar Pharmaceuticals, Inc., Rancho Cucamonga, California) in 25ml normal saline will be administered over 10 minutes. The investigators also will administer a supplementary IV infusion dose of 0.1mg/kg/hour naloxone immediately after bolus infusion will cease till the end of the experiment.
  Saline: A 0.15 mg/kg bolus dose of saline in 25ml normal saline will be administered over 10 minutes. The investigators also will administer a supplementary IV infusion dose of 0.1mg/kg/hour saline immediately after bolus infusion will cease till the end of the experiment.
  Meditation: A well-validated brief meditation-based mental training regimen [four sessions; 20 min/session] is used to teach patients to independently practice closing their eyes and take a deep breath every few minutes.
Arm/Group | Mindfulness Meditation | Non Mindfulness Meditation
Number analyzed (Participants) | 30 | 29
units on a scale
  baseline session: supine 1 | 3.60 (2.08) | 4.69 (2.25)
  baseline session: straight leg raise test 1 | 4.83 (2.21) | 5.41 (2.46)
  baseline session: supine 2 | 4.13 (2.33) | 4.76 (2.49)
  baseline session: straight leg raise test 2 | 5.15 (2.40) | 5.78 (2.81)
  saline session: supine 1 | 3.23 (2.39) | 4.62 (2.25)
  saline session: straight leg raise test 1 | 4.37 (2.28) | 5.75 (2.40)
  saline session: supine 2 | 3.90 (2.45) | 4.37 (2.28)
  saline session: straight leg raise 2 | 3.67 (2.77) | 5.32 (2.84)
  naloxone session: supine 1 | 3.30 (2.23) | 4.82 (2.34)
  naloxone session: straight leg raise 1 | 4.30 (2.52) | 6.10 (2.30)
  naloxone session: supine 2 | 3.73 (2.46) | 5.18 (2.58)
  naloxone session: straight leg raise 2 | 3.45 (2.48) | 5.52 (2.68)
Statistical Analysis 1: Comparison: Mindfulness Meditation vs Non Mindfulness Meditation; Pain ratings were collected while lying in the supine and after each straight leg rasise test (SLR 1; SLR 2). A 2 (group) X 2 (SLR 1-rest vs. SLR 2-meditation) X 2 (supine vs. SLR) X 3 (session) repeated measure mixed model ANOVA was conducted to determine if mindfulness and non-mindfulness meditation attenuate SLR induced pain through endogenous opioids. Simple effects tests tested significant main effects and interactions to test primary study hypotheses and between-group differences; Test type: Superiority; p = .05, Mixed Models Analysis

2. Secondary Outcome: Pain Catastrophizing Scale
Description: This is a 13-item questionnaire with 3 subscales assessing rumination, magnification, and helplessness in patients. A numeric value between 0 (not at all) and 4 (all the time) is provided in response to each statement. Scores on this assessment range from 0 to 52, with higher values reflecting more salient impacts of pain on one's day to day experience. The total range is from 0 - 52.
Time Frame: The Pain Catastrophizing Scale was administered at the baseline, post-intervention session 6 and session 7. Outcome measurements will compare change in Pain Catastrophizing Scale from baseline to session 7.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mindfulness Meditation: Four sessions of mindfulness-based mental training
- Non-mindfulness Meditation: Taught to take slow deep breaths across four mental training sessions.
Arm/Group | Mindfulness Meditation | Non-mindfulness Meditation
Number analyzed (Participants) | 30 | 29
units on a scale
  Baseline PCS | 18.57 (13.21) | 20.83 (12.85)
  Session 7 PCS | 15.33 (10.53) | 18.48 (13.43)

3. Secondary Outcome: The Roland-Morris Disability Questionnaire (RMDQ)
Description: The Roland-Morris Questionnaire (RMDQ) is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale. The RMDQ has been shown to yield reliable measurements, which are valid for inferring the level of disability, and to be sensitive to change over time for groups of patients with low back pain. Higher scores indicate greater disability. Total RMDQ scores are used before and after each intervention by group. The range of scores is from 0 - 24.
Time Frame: The Roland-Morris Disability Questionnaire was administered at the baseline, post-intervention session 6 and session 7. Outcome measurements will compare RMDQ from baseline to session 7.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Meditation | Non-mindfulness Meditation
Number analyzed (Participants) | 30 | 29
units on a scale
  baseline RMDQ | 12.86 (5.61) | 13.85 (6.34)
  session 7 RMDQ | 12.03 (5.71) | 14.02 (6.41)

4. Secondary Outcome: Brief Pain Inventory (BPI)
Description: Pain severity and interference: impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours or the past week. Higher scores indicate higher chronic pain. BPI severity and interference scales are used and collected before and after each intervention. Higher BPI severity indicate higher chronic pain severity. Higher BPI interference scores indicate higher chronic pain interference.The scoring scale for severity and interference range from 0 - 10, respectively.
Time Frame: Administered at the baseline, post-intervention session 6 and post-intervention session 7. Outcome measurements will compare in BPI severity and interference from baseline to session 7.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Meditation | Non-mindfulness Meditation
Number analyzed (Participants) | 30 | 29
units on a scale
  baseline BPI severity | 4.47 (1.80) | 5.22 (1.91)
  session 7 BPI severity | 3.94 (1.84) | 5.15 (2.17)
  baseline BPI interference | 4.40 (2.73) | 5.17 (2.50)
  session 7 BPI interference | 3.38 (2.34) | 4.57 (2.80)

5. Other Pre Specified Outcome: SF-12 Health Survey (SF-12) Physical Functioning
Description: This is a 12-item version of the SF-12 item Health Survey designed to assess general mental and physical functioning, and overall health-related quality of life. We used the physical functioning SF-12 scale and collected this information before and after each intervention and by group. The total range of scores is from 0 - 100. The minimum total score is 0 and the maximum score is 100. Higher scores indicate better functioning.
Time Frame: Up to 8 weeks. Administered at visit 1, 6 and 7. Outcome measurements will compare SF-12 health survey from baseline to session 7.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Meditation | Non-mindfulness Meditation
Number analyzed (Participants) | 30 | 29
units on a scale
  baseline SF physical functioning | 52.50 (28.88) | 49.17 (29.71)
  session 7 SF physical functioning | 39.66 (33.08) | 44.83 (33.66)

6. Post Hoc Outcome: Perceived Intervention Effectiveness Was Assessed With a VAS ("0" = Not Effective at All; "10" = Most Effective Imaginable) for Each Intervention Session.
Time Frame: Delivered after completion of each of the 4 meditation intervention sessions. Up to 8 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Meditation | Non-mindfulness Meditation
Number analyzed (Participants) | 30 | 29
units on a scale
  intervention 1 effectiveness | 4.83 (3.08) | 5.13 (2.63)
  intervention 2 effectiveness | 4.05 (2.45) | 5.17 (2.84)
  intervention 3 effectiveness | 4.21 (2.72) | 5.21 (2.49)
  intervention 4 effectiveness | 4.51 (2.88) | 5.40 (2.75)

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated from informed consent to data completion. This was observed in each study participant for an average of 8 weeks (i.e., through study completion).
Description: Adverse Event: any problematic medical occurrence in a subject during study participation. Adverse events were assessed in each study participant from the time of informed consent to study completion (on average of 8 weeks).
Groups:
- Mindfulness Meditation During Pain Testing, Saline and Naloxone Infusion; Non-mindfulness Meditation During Pain Testing, Saline and Naloxone Infusion: All participants were administered the straight leg raise test across all testing sessions. After their respective interventions, participants were administered the straight leg raise test during naloxone and saline infusion, respectively.
  Naloxone: A 0.15 mg/kg bolus dose of naloxone (Naloxone hydrochloride, Amphastar Pharmaceuticals, Inc., Rancho Cucamonga, California) in 25ml normal saline will be administered over 10 minutes. The investigators also will administer a supplementary IV infusion dose of 0.1mg/kg/hour naloxone immediately after bolus infusion will cease till the end of the experiment.
  Saline: A 0.15 mg/kg bolus dose of saline in 25ml normal saline will be administered over 10 minutes. The investigators also will administer a supplementary IV infusion dose of 0.1mg/kg/hour saline immediately after bolus infusion will cease till the end of the experiment.
Arm/Group | Mindfulness Meditation During Pain Testing, Saline and Naloxone Infusion | Non-mindfulness Meditation During Pain Testing, Saline and Naloxone Infusion
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 0/35 | 0/36

LIMITATIONS AND CAVEATS:
The most significant limitation was performing highly invasive pain and pharmacologic testing during the coronavirus pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT04034004/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT04034004/SAP_001.pdf
  • Informed Consent Form (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT04034004/ICF_002.pdf